CLINICAL TRIAL: NCT01340729
Title: A Phase I/II Open-Label Study of TPI 287 for Patients With Metastatic Melanoma
Brief Title: Open-Label Study of TPI 287 for Patients With Metastatic Melanoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cortice Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0839
Record Dates: First submitted 2011-04-20; First posted 2011-04-25 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; TPI 287; tumor recurrence; tumor progression; novel taxane analog
MeSH Terms: conditions — Melanoma; Recurrence; Disease Progression | interventions — TPI-287

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TPI 287 (Experimental): Starting dose TPI 287 of 125 mg/m2 intravenous (IV) for 3 weeks of 4 week schedule.
  Interventions: Drug: TPI 287

INTERVENTIONS:
Drug: TPI 287 — Starting dose of 125 mg/m2 IV via a central venous catheter (CVC) or a peripherally inserted central catheter (PICC) line over 60 minutes (+/- 10 minutes) on Days 1, 8, and 15 (+/- 2 days) of each 28 day (+/- 3 days) study cycle. The 4-week schedule composes one cycle.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of TPI 287 that can be given to patients with metastatic melanoma. Researchers want to find out if TPI 287 can control the disease. The safety of TPI 287 will also be studied.

DETAILED DESCRIPTION:
The Study Drug TPI 287 is designed to block tumors from growing by preventing cancer cells from dividing, which may cause them to die.

Study Groups:

Patient will be assigned to a study group based on when they join this study. Up to 4 groups of 3-6 participants will be enrolled in the Phase I portion of the study, and up to 64 participants will be enrolled in Phase II.

If patient is enrolled in the Phase I portion, the dose of TPI 287 they receive will depend on when they joined this study. The first group of participants will receive the lowest dose level of TPI 287. Each new group will receive a higher starting dose of TPI 287 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of TPI 287 is found.

If patient is enrolled on one of the earlier dose levels, and they do not experience intolerable side effects after 2 study cycles, their dose may be increased to the next higher dose level that has been shown to be safe.

If patient has intolerable side effects, their dose may be lowered, paused, or stopped completely. This will be up to their doctor.

If patient is enrolled in the Phase II portion, they will receive TPI 287 at the highest dose that was tolerated in the Phase I portion.

Study Drug Administration:

Each study cycle is about 28 days (+/- 3 days).

TPI 287 will be given by vein over about 1 hour, on Days 1, 8, and 15 (+/- 2 days) of each study cycle.

Since TPI 287 does not mix well in water, patient will receive doses of TPI 287 that have been dissolved in cremophor. Cremophor is a chemical that is created from castor oil. Some participants may be allergic to cremophor. Before patient receives each dose of TPI 287, they will receive dexamethasone, Benadryl (diphenhydramine), and Pepcid (famotidine) by vein, to help prevent allergic reaction. Each of these medications will be given over about 10 minutes. Patient will also receive drugs to prevent nausea and vomiting. The study staff will tell patient more about these drugs and the risks for them.

Study Visits:

At all study visits, patient will be asked about any symptoms they may be having and any drugs they may be taking.

On Days 1, 8, 15, and 21 of each cycle, blood (about 1 teaspoon) will be drawn for routine tests. The blood sample on Day 21 may be drawn at a clinic near patient's home. The study staff will give patient more information about this.

On Day 28 of each cycle:

* Patient will have a physical exam, including measurement of their height, weight, and vital signs.
* Patient's performance status will be recorded.
* Blood (about 1 teaspoon) will be drawn for routine tests.
* If the doctor thinks it is needed, patient will have an MRI scan of the brain to check the status of the disease.
* If the doctor thinks it is needed, patient will have a neurological exam.

On Day 1 of Cycle 2 and then every other cycle after that (Cycles 2, 4, 6, and so on), patient will have a CT scan of their chest, abdomen, and pelvis to check the status of the disease.

Every 8 weeks, patient will have a CT or MRI scan of the brain to check the status of the disease. If patient has brain metastasis, they will have a CT or MRI scan every 4 weeks.

Length of Study:

Patient may continue taking the study drug for up to 6 months. Treatment beyond 6 months will be decided by patient's doctor. Patient will be allowed to continue taking the study drug for as long as the doctor thinks it is in their best interest. Patient will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation on the study will be over once they have completed the end-of-treatment visit and follow-up.

End-of-Treatment Visit:

About 4 weeks after patient stops receiving TPI 287, they will have an end-of-treatment visit. At this visit, the following tests and procedures will be performed:

* Patient will have a physical exam, including measurement of their weight and vital signs.
* Patient's performance status will be recorded.
* Patient will be asked about any problems or side effects they may be having.
* Blood (about 2 tablespoons) will be drawn for routine tests.
* If patient's doctor thinks it is needed, they will have a CT or MRI scan to check the status of the disease.

Follow-Up:

* Patient will be contacted by phone or they will come in for a clinic visit. The phone call should last about 5 minutes. Patient will be asked about any problems or side effects they may be having:
* Every 2 months unless the disease gets worse.
* Then, every 3 months after that.

These follow-ups end 3 years after they enrolled in the study.

This is an investigational study. TPI 287 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 82 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven melanoma with metastasis that is unresectable Stage III or Stage IV. This will include bulky stage III and M1-3.
2. Patients must have shown unequivocal evidence for tumor recurrence or progression and should have at least one indicator lesion that can be measured in one dimension as >/= 20mm with conventional techniques (CT, MRI, and X-ray) or >/= 10mm with spiral CT scan.
3. Patients with melanoma with documented metastases to the brain are eligible: a. Must be asymptomatic with stable disease for at least 2 months as determined by CT or MRI of the brain at the time of evaluation no measurable changes. b. May have had prior therapy for brain metastasis such as whole brain irradiation, stereotactic gamma ray therapy or resection of brain metastases.
4. Patients may have had up to two prior cytotoxic chemotherapy regimens for their systemic disease (immunological or targeted therapy e.g. vaccine, IL-2, B-RAF inhibitors, will not be considered prior cytotoxic chemotherapy)
5. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital.
6. Patients must have a Eastern Cooperative Oncology Group (ECOG) status of </= 2.
7. Patients must have recovered from the toxic effects of prior therapy (baseline grade), at least 3 weeks after the last dose was administered. Any questions about whether patients fulfill this criteria should be directed to the Study Chair.
8. Patients must have adequate bone marrow function (Absolute neutrophil count (ANC)>/= 1,500/mm^3 and platelet count of >/= 100,000/mm^3), adequate liver function [aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT or SGPT) </= 2.5 times normal for patients without liver metastasis and ALT (SGPT) and AST (SGOT) </= 5, times normal for patients with liver metastasis], serum bilirubin </= 2 mg/dl), and adequate renal function (BUN and creatinine >/= 1.5 times institutional normal) prior to starting therapy
9. As TPI 287 may interfere with Coumadin dosing, patients who are taking TPI 287 will require monitoring of their Prothrombin Time (PT), Partial thromboplastin time (PTT) and International Normalized Ratio (INR)
10. Females of childbearing potential (non childbearing is defined as greater than one year post-menopausal or surgically sterilized) must use acceptable contraceptive methods (abstinence, intrauterine device, oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this trial. Sexually active men must also use acceptable contraceptive methods for the duration of time on study.
11. Patient should be 15 years of age or older

Exclusion Criteria:

1. 1. Patients with brain metastases not stable for 2 months.
2. Patients taking primidone, carbamazepine, phenobarbital or phenytoin anticonvulsants (Enzyme-Inducing Anti-Epileptic Drugs - EIAED). Patients changing from these anticonvulsants to others that are allowed must be off the drugs listed above for at least 1 week before start of treatment.
3. Patients with > Grade 2 neuropathy
4. Patients with uncontrolled high blood pressure (systolic BP > 140 for patients < 50 years old and >160 for patients > 50 and/or diastolic BP>90 for patients< 50 year old and >99 for patients over 50) unstable angina, symptomatic congestive heart failure, clinical history of myocardial infarction within the previous six months, or serious uncontrolled cardiac arrhythmia as determined by the principal investigator.
5. Because of the concerns for the potential interaction of TPI 287 and medications taken by patients who are HIV positive or have AIDS related diseases, patients who are HIV positive are not eligible for entry into this study. Only patients with suspected HIV will be tested and if positive, will be ineligible.
6. Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) are ineligible unless in complete remission and off of all therapy for that disease for a minimum of 3 years.
7. Patients with: a. Active infection associated with fever lasting more than 24 hours requiring antibiotics b. Disease that will obscure toxicity or dangerously alter drug metabolism c. Serious intercurrent medical illness The Principal investigator or his designee will make the final decision regarding eligibility for enrollment.
8. Female patients who are pregnant or breastfeeding
9. Patients younger than 15 years of age

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) TPI 287 administered weekly for three weeks out of every four in patients with metastatic melanoma | With each 28 day cycle and DLTs at 12 weeks
  Optimal dose (MTD) of TPI 287 for the Phase II part of the study defined as level at which no dose limiting toxicities (DLTs) are experienced (3+3 dose escalation algorithm). DLT is defined as Grade 3 or higher toxicity that is reasonably likely to be associated with study treatment at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Agop Y. Bedikian, MD, BS, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org